CLINICAL TRIAL: NCT01306058
Title: A Phase I/II Study of TRC105 in Combination With Sorafenib in Hepatocellular Carcinoma (HCC)
Brief Title: Sorafenib and TRC105 in Hepatocellular Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Tim Greten, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110102; 11-C-0102
Record Dates: First submitted 2011-02-26; First posted 2011-03-01 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Hepatoma; Liver Neoplasms; Adenoma, Liver Cell; Carcinoma, Hepatocellular; Liver Neoplasms, Experimental
Keywords: Hepatocellular Carcinoma; TRC105; Sorafenib; Liver Cancer; Monoclonal Antibody
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms; Adenoma, Liver Cell; Liver Neoplasms, Experimental | interventions — carotuximab; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sorafenib & TRC105 in Hepatocellular CA (Experimental): CA (cancer); 15 mg/kg TRC105 intravenous (IV) every 2 weeks and 400 mg sorafenib by mouth (PO) twice per day
  Interventions: Drug: TRC 105; Drug: Sorafenib

INTERVENTIONS:
Drug: TRC 105 — 15 mg/kg intravenous (IV) every 2 weeks
Drug: Sorafenib — 400 mg twice a day (bid) continuously in a 28 days cycle
  Other Names: Nexavar

SUMMARY:
Background:

Sorafenib is a drug that has been approved to treat kidney and liver cancer (hepatocellular carcinoma, or HCC) and has been shown to prolong survival in patients with HCC. It works by slowing the spread of cancer cells, but it does not fully prevent the cancer from growing again. Researchers are interested in combining sorafenib with the experimental drug TRC105, which has been designed to block the growth of blood vessels that lead to tumor growth, in order to determine whether this drug combination stops tumor growth and reduces tumor size better than sorafenib alone.

Objectives:

To determine the safety and effectiveness of the combination of sorafenib and TRC105 as a treatment for hepatocellular cancer that has not responded to other treatments.

Eligibility:

Individuals at least 18 years of age who have been diagnosed with hepatocellular cancer that has not responded to other treatments, and who are not considered to be candidates for liver transplantation. Patients cannot be receiving anticoagulant therapy with the exception of low dose aspirin. No history of bleeding problems or peptic ulcer disease.

Design:

Participants will be screened with a full medical history and physical examination, blood and urine tests, and tumor imaging studies. Participants will have a tumor biopsy or provide previously collected tumor tissue for study. An examination of the esophagus to look for problems with blood vessels will be completed in patients with a history of cirrhosis.

Participants will receive sorafenib tablets twice every day, in the morning and at night, with a full glass of water.

Participants will receive TRC 105 infusions once every two weeks on days 1 and 15 of a 28 day cycle.

At each visit during the first cycle, participants will have a physical examination and blood tests. Participants will continue to have blood tests and a urine test every cycle to monitor the effects of treatment, including tests of kidney function. Participants will have imaging studies after every two cycles to evaluate the results of treatment, and may also provide tumor samples for study.

Treatment will continue as long as the tumor does not grow and side effects remain tolerable.

DETAILED DESCRIPTION:
Background:

* Worldwide, hepatocellular carcinoma (HCC) is the fifth most common malignancy with a median survival of 6-9 months. The Study of Heart and Renal Protection (SHARP) study established sorafenib as a standard consideration in this disease and set the bar for future studies of systemic therapy.
* TRC105 is a chimeric anti-angiogenic monoclonal antibody that binds cluster of differentiation 105 (CD105), a transmembrane receptor selectively expressed by proliferating endothelial cells. TRC105 binds to CD105-expressing endothelial cells and mediates growth inhibition, apoptosis and antibody-dependent cell-mediated cytotoxicity (ADCC).

Objectives:

Primary:

* Phase I: To establish the maximum tolerated dose (MTD) of TRC105 when given with standard-dose sorafenib for HCC.
* Phase II:To determine the estimate response rate according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria for the combination of TRC105 with sorafenib in HCC.

Eligibility:

* Histologically or cytologically confirmed diagnosis of HCC.
* Childs-Pugh A or B (7 points) cirrhosis is allowed.
* Patients must have disease that is not amenable to potentially curative resection, radiofrequency ablation, or liver transplantation.
* In phase I, prior systemic therapy is allowed.
* In phase II, prior systemic therapy for HCC (including sorafenib) is allowed.
* No history of bleeding varices in previous 1 year (unless subsequent liver transplant).
* No anti-coagulation (except low-dose aspirin).

Design:

* TRC105 will be administered intravenously every two weeks, on days 1 and 15 of each 28 day cycle. Sorafenib will be self-administered twice daily by mouth.
* Phase 1: The first part of this study was a standard 3+3 dose escalation phase I study with the primary objective of establishing MTD for TRC105 when given in combination with standard-dose sorafenib. Sorafenib is taken orally at a dose of 400 mg twice daily. TRC105 is administered as an intravenous infusion every two weeks. Patients will be restaged including imaging studies to assess for response and progression every 8 weeks. The TRC105 dose was escalated in cohorts of 3 to 6 patients up to a maximum of 15 mg/kg every two weeks. Intra-patient dose escalation was not allowed.
* Phase II: TRC105 will be administered as an intravenous infusion every two weeks at the recommended phase II dose, 15 mg/kg of TRC105 ever two weeks in combination with standard dose sorafenib, defined in phase I. The sample size and interim stopping rule will be determined using a Simon optimal two-stage design. The first stage will initially enroll 6 evaluable patients, and if 0 of the 6 have a clinical response, then no further patients will be accrued. If 1 or more of the first 6 patients has a clinical response, then accrual would continue until a total of 23 patients have been enrolled. As it may take several weeks to determine if a patient has experienced a response, a temporary pause in the accrual may be necessary to ensure that enrollment to the second stage is warranted. If there are 1 to 2 clinical responses in 23 patients, this would be an uninterestingly low response rate. If there were 3 or more complete responses in 23 patients (13.0%), this would be sufficiently interesting to warrant further study in later trials. Under the null hypothesis (5% response rate), the probability of early termination is 73.5%.

Cohort: -0; Sorafenib (mg by mouth (PO) twice daily): 400 bid; TRC105 (mg/kg intravenous (IV) weekly): 1

Cohort: 1; Sorafenib (mg PO twice daily): 400 bid; TRC105 (mg/kg IV weekly): 3

Cohort: 2; Sorafenib (mg PO twice daily): 400 bid; TRC105 (mg/kg IV weekly): 6

Cohort: 3; Sorafenib (mg PO twice daily): 400 bid; TRC105 (mg/kg IV weekly): 10

Cohort: 4; Sorafenib (mg PO twice daily): 400 bid; TRC105 (mg/kg IV weekly): 15

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histopathological confirmation of hepatocellular carcinoma (HCC) by the Laboratory of Pathology of the National Cancer Institute (NCI) prior to entering this study.

Or

histopathological confirmation of carcinoma in the setting of clinical and radiological characteristics which, together with the pathology, are highly suggestive of a diagnosis of HCC.

* Patients must have disease that is not amenable to potentially curative resection or ablative techniques. In addition, disease must not be amenable to or have progressed on transhepatic arterial chemoembolization (TACE). Patients must not be considered potential candidates for liver transplantation. This determination will be made after hepatobiliary surgical input at the NCI multidisciplinary conference.
* If liver cirrhosis is present, patient must have a Child-Pugh A classification.
* Patients with cirrhosis must have had esophagogastric endoscopy within the previous 6 months prior to study entry for the assessment of varices. If the patient has not had this done they must be willing to undergo this procedure prior to study entry.
* Age greater than or equal to 18 years
* Life expectancy of greater than 3 months.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Patients must have normal organ and marrow function as defined below:

  * Absolute neutrophil count greater than or equal to 1,500/mcL
  * Platelets greater than or equal to 60,000/mcL without transfusion support within the past 30 days
  * Total bilirubin less than or equal to 3 mg/dl.
  * Aspartate aminotransaminase (AST)/alanine aminotransaminase (ALT) less than or equal to 10 times upper limit of normal
  * Creatinine less than or equal to 1.5 times upper normal limits OR creatinine clearance greater than or equal to 40mL/min/1.73 m^2 for patients with creatinine levels above institutional normal, as calculated by the Cockcroft Gault formula.
* Patients must have recovered from any acute toxicity related to prior therapy, including surgery. Toxicity should be less than or equal to grade 1 or returned to baseline.
* Patients must not have other invasive malignancies within the past 5 years (with the exception of non-melanoma skin cancers or non-invasive bladder cancer).
* Patient must be able to understand and willing to sign a written informed consent document.

Additional Inclusion Criteria for PHASE I Portion:

* Patients may have measurable or evaluable disease only.
* Prior therapy: prior systemic therapy with sorafenib is allowed.

Additional Inclusion Criteria for PHASE II Portion:

* All patients will be required to have measurable disease.
* Prior therapy: prior systemic therapy with sorafenib is allowed.

EXCLUSION CRITERIA:

* Patients who have had chemotherapy (other than sorafenib treatment), large field radiotherapy, or major surgery must wait 4 weeks prior to entering the study.
* Patients may not be receiving any agents not approved by the Food and Drug Administration (FDA) within the past 4 weeks.
* Patients with known brain metastases will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Proteinuria, as demonstrated by a 24-hour protein of greater than or equal to 2000 mg. Urine protein will be screened by urine protein-creatinine ratio (UPC). For UPC ratio greater than 1.0, a 24-hour urine protein will need to be obtained and the level should be less than 2000 mg for patient enrollment.
* Uncontrolled intercurrent illness including, but not limited to, hypertension (systolic blood pressure (BP) greater than 140, diastolic BP greater than 90), ongoing or active systemic infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia or psychiatric illness/social situations that would limit compliance with study requirements.
* No anti-coagulation therapy is allowed with the exception of low-dose aspirin.
* No bleeding diathesis.
* Patients with a history of bleeding varices in previous 1 year are excluded (unless patient has subsequently had a liver transplant. Those with gastric varices or varices that are deemed as high risk by the endoscopist should be placed on appropriate medical therapy as advised by the gastroenterologist.
* History of peptic ulcer disease or gastritis within 6 months of TRC105 administration, unless patient has received adequate treatment for peptic ulcer disease and has evidence of complete resolution documented by esophagogastroduodenoscopy (EGD). Mild gastritis is allowed.
* Corrected QT interval (QTc) greater than 500 msec
* Human immunodeficiency virus (HIV)-positive patients receiving anti-retroviral therapy are excluded from this study due to the possibility of pharmacokinetic interactions between antiretroviral medications and sorafenib or TRC105. HIV positive patients not receiving antiretroviral therapy are excluded due to the possibility that sorafenib or TRC105 may worsen their condition and the likelihood that the underlying condition may obscure the attribution of adverse events with respect to sorafenib or TRC105.
* History of hypersensitivity reaction to human or mouse antibody products
* Patients with a history of familial bleeding disorders
* Patients with a history of hereditary hemorrhagic telangiectasia (Osler-Weber- Rendu Syndrome).
* Pregnancy and breast feeding are exclusion factors. Enrolled patients must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, the duration of study participation and 3 months after the end of the treatment.
* Patients with unhealed wounds for more than 30 days.

INCLUSION OF WOMEN AND MINORITIES:

-Men and women of all races and ethnic groups are eligible for this trial.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-02-11 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2017-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim F Greten, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Parkin DM, Bray F, Ferlay J, Pisani P. Estimating the world cancer burden: Globocan 2000. Int J Cancer. 2001 Oct 15;94(2):153-6. doi: 10.1002/ijc.1440. No abstract available. PMID 11668491
- [Background] Yoo HY, Patt CH, Geschwind JF, Thuluvath PJ. The outcome of liver transplantation in patients with hepatocellular carcinoma in the United States between 1988 and 2001: 5-year survival has improved significantly with time. J Clin Oncol. 2003 Dec 1;21(23):4329-35. doi: 10.1200/JCO.2003.11.137. Epub 2003 Oct 27. PMID 14581446
- [Background] Palmer DH. Sorafenib in advanced hepatocellular carcinoma. N Engl J Med. 2008 Dec 4;359(23):2498; author reply 2498-9. No abstract available. PMID 19065750
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-C-0102.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 27 patients were enrolled. One patient signed consent but developed rapid disease progression and did not receive any treatment.
Groups:
- Sorafenib & TRC105 in Hepatocellular CA: CA (cancer); 15 mg/kg TRC105 intravenous (IV) every 2 weeks and 400 mg sorafenib by mouth (PO) twice per day
  TRC 105: 15 mg/kg IV every 2 weeks
  Sorafenib: 400 mg twice a day (bid) continuously in a 28 days cycle
Period: Overall Study
Arm/Group | Sorafenib & TRC105 in Hepatocellular CA
Started | 27
Completed | 25
Not Completed | 2
Not completed — Death | 1
Not completed — Enrolled but did not get treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sorafenib & TRC105 in Hepatocellular CA
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 13
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27
Participant Etiology of Hepatocellular Cancer (HCC) [Count of Participants; unit: Participants] — Hepatitis B virus is a viral infection that affects the liver. Hepatitis C virus is a virus spread by infected blood (e.g. share needles). Crytogenic means the cause of the disease is unknown. Hematochromatosis is an iron disorder in which the body has an excess of iron in the blood. Population: One patient was enrolled and signed consent but developed rapid disease progression and did not receive any treatment. One patient developed a fatal myocardial infarction.
  Participants
    Hepatitis B Virus (HBV): number analyzed (Participants) | 25
    Hepatitis B Virus (HBV) | 3
    Hepatitis C Virus (HCV): number analyzed (Participants) | 25
    Hepatitis C Virus (HCV) | 15
    Cryptogenic: number analyzed (Participants) | 25
    Cryptogenic | 6
    Hematochromatosis: number analyzed (Participants) | 25
    Hematochromatosis | 1
Baseline Child Pugh Score [Count of Participants; unit: Participants] — The Modified Child-Pugh classifies the severity of liver disease according to the degree of ascites, plasma concentrations of bilirubin and albumin, the prothrombin time and degree of encephalopathy. A total score of 5-6 is considered grade A (well-compensated disease); 7-9 grade B (significant functional compromise) and 10-15 is grade C (decompensated disease). NA = not all patients had cirrhosis. You only do a Pugh Score if cirrhosis is present. Population: One patient was enrolled and signed consent but developed rapid disease progression and did not receive any treatment. One patient developed a fatal myocardial infarction.
  Participants
    Child Pugh Score - 5: number analyzed (Participants) | 25
    Child Pugh Score - 5 | 10
    Child Pugh Score - 6: number analyzed (Participants) | 25
    Child Pugh Score - 6 | 4
    Child Pugh Score - 7: number analyzed (Participants) | 25
    Child Pugh Score - 7 | 1
    NA: number analyzed (Participants) | 25
    NA | 10
Number of Participants with Extrahepatic disease [Count of Participants; unit: Participants] — Extrahepatic is defined as disease outside of the liver. Population: One patient was enrolled and signed consent but developed rapid disease progression and did not receive any treatment. One patient developed a fatal myocardial infarction.
  Participants
    Yes: number analyzed (Participants) | 25
    Yes | 17
    No: number analyzed (Participants) | 25
    No | 8
Prior Therapies [Count of Participants; unit: Participants] — Of note, some patients received more than one prior therapeutic intervention. Transcatheter arterial chemoembolization (TACE) is performed to restrict blood flow. Ablation is a procedure to destroy cardiac tissue. Radioembolization is a combination of embolization and radiation therapy to treat liver cancer. Locoregional is a recurrence of cancer at the same original site of disease. Transplant refers to a liver transplant.
  Participants
    No prior intervention | 9
    ≥2 locoregional procedures | 7
    Previous TACE | 8
    Surgery | 5
    Ablation | 2
    Radioembolization | 2
    Transplant | 2
Number of Participants with Liver Cirrhosis [Count of Participants; unit: Participants] — Cirrhosis is scar tissue on the liver. Population: One patient was enrolled and signed consent but developed rapid disease progression and did not receive any treatment. One patient developed a fatal myocardial infarction.
  Participants
    Yes: number analyzed (Participants) | 25
    Yes | 15
    No: number analyzed (Participants) | 25
    No | 10
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG Grade 0 is normal activity. Fully active, able to carry on all-pre-disease performance without restriction. Grade 1 is symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature. Grade 2 is in bed <50% of the time. Ambulatory and capable of all self-care, but unable to carry out any work activities. Grade 3 is in bed >50% of the time. Capable of only limited self-care, confined to bed or chair more than 50% of waking hours. Grade 4 is 100% bedridden. Completely disabled. Grade 5 is dead. Population: One patient was enrolled and signed consent but developed rapid disease progression and did not receive any treatment. One patient developed a fatal myocardial infarction.
  Participants
    Grade 0: number analyzed (Participants) | 25
    Grade 0 | 8
    Grade 1: number analyzed (Participants) | 25
    Grade 1 | 17
Participants with Hepatocellular Cancer & Fibrolamellar [Count of Participants; unit: Participants] — HCC is liver cancer usually found in patients with cirrhosis or liver disease. Fibolamellar is a rare form of HCC. The tumor cells are mixed with fibrous layers. Population: One patient was enrolled and signed consent but developed rapid disease progression and did not receive any treatment. One patient developed a fatal myocardial infarction.
  Participants
    Hepatocellular Cancer (HCC): number analyzed (Participants) | 25
    Hepatocellular Cancer (HCC) | 24
    Fibrolamellar: number analyzed (Participants) | 25
    Fibrolamellar | 1

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Maximum Tolerated Dose (MTD) of TRC105 When Given With Standard-dose Sorafenib for Hepatocellular Cancer (HCC)
Description: MTD is the highest dose studied for which the incidence of DLT was less than 33%. DLT criteria included treatment-related grade 3 non-hematological toxicities or grade 4 hematological toxicities occurring within the first 28 days of treatment. Grade 3 electrolyte toxicities to be corrected to Grade 1 or less within 24 hours will be considered dose limiting (proteinuria >3.5g/24 hour will be defined as a DLT). Drug-related Grade 4 hematological toxicity will be considered dose limiting. Toxicity requiring a dose reduction or a delay in treatment for >7 days will be considered dose limiting. Other Grade 3 or higher toxicity related to TRC105 will be considered dose limiting.
Time Frame: Completed in the first 28 days of treatment (cycle 1)
Population: 24/27 analyzed. One patient signed consent but developed rapid disease progression and did not receive any treatment. One patient developed a fatal myocardial infarction and one patient developed a grade 3 cerebral tumor hemorrhage.
Measure: Number; unit: mg/kg
Arm/Group | Sorafenib & TRC105 in Hepatocellular CA
Number analyzed (Participants) | 24
mg/kg | 15

2. Primary Outcome: Phase II: Time to Progression (TTP) for the Combination of TR105 With Sorafenib in Hepatocellular Cancer (HCC)
Description: TTP is the time between the first day of treatment to the day of disease progression. Progressive disease was measured by the Response Evaluation Criteria in Solid Tumors (RECIST) and is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. (Note: the appearance of one or more new lesions is also considered progressions).
Time Frame: 2 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sorafenib & TRC105 in Hepatocellular CA
Number analyzed (Participants) | 24
Months | 3.8 [3.2 to 5.6]

3. Secondary Outcome: Overall Response Rate (ORR) as Determined by the Standard Response Evaluation Criteria in Solid Tumors (RECIST) Criteria
Description: Overall response (Complete Response (CR) + Partial Response (PR) was assessed by the Standard Response Evaluation Criteria in Solid Tumors (RECIST) criteria for target lesions and assessed by magnetic resonance imaging (MRI). CR is disappearance of all target lesions. PR is at least a 30% decrease in the sum of the longest diameter of target lesions.
Time Frame: 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sorafenib & TRC105 in Hepatocellular CA
Number analyzed (Participants) | 24
percentage of participants | 21 [7.1 to 42.2]

4. Secondary Outcome: Overall Response Rate (ORR) as Determined by the European Association for the Study of the Liver (EASL)-Modified Response Evaluation Criteria in Solid Tumors (RECIST) Criteria
Description: Overall response (Complete Response (CR) + Partial Response (PR) was assessed by the European Association for the Study of the Liver (EASL)-modified Response Evaluation Criteria in Solid Tumors (RECIST) criteria for target lesions and assessed by magnetic resonance imaging (MRI). CR is disappearance of all target lesions. PR is at least a 30% decrease in the sum of the longest diameter of target lesions.
Time Frame: 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sorafenib & TRC105 in Hepatocellular CA
Number analyzed (Participants) | 24
percentage of participants | 21 [7.1 to 42.2]

5. Secondary Outcome: Patients Who Developed Antidrug Antibodies
Description: Patients who develop antidrug antibodies is measured by human anti-chimeric antibody (HACA) formation (e.g. immunogenicity of TRC105).
Time Frame: Cycle 1 Day 1, 28 days post end of study (up to 2 years)
Population: 11/27 were analyzed because only 11 patients were evaluable at the highest dose level given to patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib & TRC105 in Hepatocellular CA
Number analyzed (Participants) | 11
Participants | 7

6. Secondary Outcome: Immunogenicity of TRC105 as Measured by Human Anti-mouse Antibody (HAMA) Formation
Description: A 5mL blood sample will be collected to assess immunogenicity. Immunogenicity will be measured by the enzyme-linked immunosorbent assay (ELISA) and expressed in titres. The higher the titre, the higher the formation of HAMA antibody in the blood. A higher concentration of HAMA (higher titre result) is a negative finding. A higher level means the drug elimination is faster and the TRC 105 is then less effective. Lower level is 0-2 titre. Any value above 2 titre would be a positive HAMA result. The HAMA ( Human anti-mouse antibody) measurement at 28 days post treatment levels provides information as to the rate of drug elimination and effectiveness. Patients with 0 to < 2.0 titre. eliminates the TRC 105 slower and the drug may be more effective than patients who have a low(>2.0 titres) or high level of HAMA. Higher levels of HAMA reflect the TRC 105 elimination from the body faster and the drug potentially not as effective as negative HAMA titres.
Time Frame: Baseline and then 28 days following the end of the study treatment, approximately two years
Population: 9/20, 8/20, and 3/20 participants were evaluable for the noted time periods below.
Measure: Geometric Mean (95% Confidence Interval); unit: titres
Arm/Group | Sorafenib & TRC105 in Hepatocellular CA
Number analyzed (Participants) | 20
titres
  Baseline | 0.02 [0 to 2]
  no evidence of HAMA 28 days post treatment: number analyzed (Participants) | 9
  no evidence of HAMA 28 days post treatment | 0 [0 to 0]
  Low level of HAMA 28 days post treatment: number analyzed (Participants) | 8
  Low level of HAMA 28 days post treatment | 65 [2 to 128]
  High level of HAMA 28 days post treatment: number analyzed (Participants) | 3
  High level of HAMA 28 days post treatment | 515 [256 to 1024]

7. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events by Common Terminology Criteria in Adverse Events (CTCAE)v4.0
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: 4 years and 10.5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib & TRC105 in Hepatocellular CA
Number analyzed (Participants) | 27
Participants | 27

8. Secondary Outcome: Number of Participants With Dose Limiting Toxicity (DLT)
Description: DLT was assessed by the Common Terminology Criteria in Adverse Events (CTCAE) v4.0. DLT criteria included treatment-related grade 3 non-hematological toxicities or grade 4 hematological toxicities occurring within the first 28 days of treatment. Grade 3 electrolyte toxicities to be corrected to Grade 1 or less within 24 hours will be considered dose limiting (proteinuria >3.5g/24 hour will be defined as a DLT). Drug-related Grade 4 hematological toxicity will be considered dose limiting. Toxicity requiring a dose reduction or a delay in treatment for >7 days will be considered dose limiting. Other Grade 3 or higher toxicity related to TRC105 will be considered dose limiting.
Time Frame: First 28 days of treatment (cycle 1)
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib & TRC105 in Hepatocellular CA
Number analyzed (Participants) | 27
Participants | 1

9. Secondary Outcome: Treatment-emergent Adverse Events
Description: Here are the number of treatment-emergent adverse events categorized by Any grade, Grade 3, Grade 4 and Grade 5 adverse events. Adverse events was assessed by the Common Terminology Criteria in Adverse Events (CTCAE) v4.0. Grade 1 is mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 is moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL) (e.g. preparing meals, shopping for groceries or clothes). Grade 3 is severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL (e.g. bathing, dressing and undressing). Grade 4 is life-threatening consequences; urgent intervention indicated. Grade 5 is death related to adverse event.
Time Frame: 4 years and 10.5 months
Population: 25/27 analyzed. One patient developed a fatal myocardial infarction and one patient developed a grade 3 cerebral tumor hemorrhage.
Measure: Number; unit: treatment-emergent adverse events
Arm/Group | Sorafenib & TRC105 in Hepatocellular CA
Number analyzed (Participants) | 25
treatment-emergent adverse events
  Any Grade Headache | 20
  Any Grade Epistaxis | 19
  Any Grade Increased aspartate aminotransaminase | 18
  Grade 3 Increased aspartate aminotransaminase | 5
  Any Grade Rash, other | 18
  Grade 3 Rash, other | 3
  Any Grade Hypophosphatemia | 18
  Grade 3 Hypophosphatemia | 7
  Any Grade Hypoalbuminemia | 17
  Grade 3 Hypoalbuminemia | 2
  Any Grade Anemia | 16
  Grade 3 Anemia | 1
  Any Grade Fatigue | 15
  Any Grade Increased alkaline phosphatase | 15
  Grade 3 Increased alkaline phosphatase | 5
  Any Grade Diarrhea | 15
  Grade 3 Diarrhea | 1
  Any Grade Increased blood bilirubin | 14
  Grade 3 Increased blood bilirubin | 6
  Grade 4 Increased blood bilirubin | 1
  Any Grade Nausea | 14
  Any Grade Increased alanine transaminase | 13
  Any Grade Oral mucositis/pain | 12
  Any Grade Thrombocytopenia | 10
  Grade 3 Thrombocytopenia | 1
  Any Grade Amylase | 10
  Grade 3 Amylase | 2
  Grade 4 Amylase | 1
  Any Grade Abdominal pain | 9
  Any Grade Hand-foot skin reaction | 8
  Grade 3 Hand-foot skin reaction | 2
  Any Grade Infusion reaction | 8
  Grade 3 infusion reaction | 1
  Any Grade Neutropenia | 8
  Any Grade Weight loss | 8
  Any Grade Hypertension | 6
  Grade 3 Hypertension | 1
  Any Grade Vomiting | 6
  Any Grade Hypomagnesemia | 5
  Any Grade Alopecia | 5
  Any Grade Insomnia | 4
  Any Grade Constipation | 3
  Grade 3 Intracranial hemorrhage | 1
  Grade 5 Myocardial ischemia | 1
  Grade 4 Lipase | 1
  Any Grade Hyperglycemia | 1
  Grade 3 Hyperglycemia | 2
  Grade 4 Hyperuricemia | 2

10. Secondary Outcome: Median Progression-free Survival (PFS)
Description: PFS was calculated from the on-study date until date of progression, death, or an event that would render the patient inevaluable for further follow-up (liver dysfunction), or end of study. Probabilities were determined using the Kaplan-Meier method. Progressive disease was measured by the Response Evaluation Criteria in Solid Tumors (RECIST) and is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. (Note: the appearance of one or more new lesions is also considered progressions).
Time Frame: up to 6 months
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sorafenib & TRC105 in Hepatocellular CA
Number analyzed (Participants) | 25
Months | 3.8 [3.2 to 5.6]

11. Secondary Outcome: Percentage of Participants With Progression Free Survival (PFS) at 3 and 6 Months
Description: Percentage of participants who were progression free at 3 and 6 months. Progressive disease was measured by the Response Evaluation Criteria in Solid Tumors (RECIST) and is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. (Note: the appearance of one or more new lesions is also considered progressions).
Time Frame: 3 and 6 months
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sorafenib & TRC105 in Hepatocellular CA
Number analyzed (Participants) | 25
percentage of participants
  3 month PFS | 75.0 [52.6 to 87.9]
  6 month PFS | 16.7 [5.2 to 33.7]

12. Secondary Outcome: Median Overall Survival (OS)
Description: OS was calculated from the on-study date until the date of death or the date the patient was last known to be alive. Probabilities were determined using the Kaplan-Meier method.
Time Frame: up to 2 years
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sorafenib & TRC105 in Hepatocellular CA
Number analyzed (Participants) | 25
Months | 15.5 [8.5 to 26.3]

13. Secondary Outcome: Percentage of Participants With Overall Survival (OS) at 6 and 12 Months
Description: Percentage of participants last known to be alive at 6 and 12 months.
Time Frame: 6 and 12 months
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sorafenib & TRC105 in Hepatocellular CA
Number analyzed (Participants) | 25
percentage of participants
  6 month OS | 74.0 [50.9 to 87.4]
  12 month OS | 59.2 [35.9 to 76.4]

14. Secondary Outcome: Number of Participants With Stable Disease, Partial Response, and Progressive Disease on Phase I and Phase II of the Clinical Trial
Description: Response is defined as per the Response Evaluation Criteria in Solid Tumors (RECIST). Partial response (PR) is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. To be assigned a confirmed PR, changes in tumor measurements must be confirmed by repeat assessments that should be performed at least 4 weeks after the criteria for response are first met. Stable disease is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum of diameters on study. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. (Note: the appearance of one or more new lesions is also considered progressions).
Time Frame: Every 8 weeks, up to 180 days
Population: 7/27 participants were not evaluable (1 was not evaluable, 1 patient had dose limiting toxicity myocardial infarction, 1 could not tolerate sorafenib, 1 infusion reaction to TRC105 during first dose, 1 early progressive disease, 1 side effects, and 1 off due to severe skin toxicity).
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib & TRC105 in Hepatocellular CA
Number analyzed (Participants) | 20
Participants
  Phase I - Stable disease: number analyzed (Participants) | 14
  Phase I - Stable disease | 9
  Phase I - Progressive disease: number analyzed (Participants) | 7
  Phase I - Progressive disease | 2
  Phase I - Partial response: number analyzed (Participants) | 9
  Phase I - Partial response | 4
  Phase 2 - Stable disease: number analyzed (Participants) | 6
  Phase 2 - Stable disease | 3
  Phase 2 - Partial response: number analyzed (Participants) | 6
  Phase 2 - Partial response | 1
  Phase 2 - Progressive disease: number analyzed (Participants) | 6
  Phase 2 - Progressive disease | 2

15. Secondary Outcome: Area Under the Plasma Concentration
Description: Mean peak TRC105 serum trough concentrations were plotted over time by dose level to assess accumulation. (e.g. drug absorption). The lower limit of quantification (LLOQ) is 200 ng/mL.
Time Frame: Cycle 1 Day 1, Cycle 1 Day 15, Cycle 2 Day 1, Cycle 2 Day 15, and prior to start of TRC105 infusion
Population: as for outcome 1
Measure: Mean (Full Range); unit: Hr*ng/mL
Arm/Group | Sorafenib & TRC105 in Hepatocellular CA
Number analyzed (Participants) | 24
Hr*ng/mL
  Dose level 1 | 75933 [73054 to 78813]
  Dose level 2 | 152900 [123166 to 182634]
  Dose level 3 | 242882 [196241 to 289524]
  Dose level 4 | 362611 [324921 to 400301]

16. Secondary Outcome: Changes in Biomarkers Vascular Endothelial Growth Factor (VEGF) and Placenta Growth Factor (PIGF)
Description: Plasma biomarker tests were performed for VEGF and PIGF using assay plates from Meso-Scale Discovery according to the product manual. The concentrations of the cytokines were determined with recombinant standards. Changes in biomarkers were determined by a Wilcoxon signed rank test.
Time Frame: Cycle 1 day 1, cycle 1 day 15, cycle 2 day 1, or end of study, an average of 12 weeks
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Sorafenib & TRC105 in Hepatocellular CA
Number analyzed (Participants) | 25
pg/ml
  VEGF cycle 1 day 1 | 202.5 [100.9 to 341.5]
  PIGF cycle 1 day 1 | 44.6 [39.9 to 54.1]
  VEGF cycle 1 day 15 | 299 [149.2 to 520.5]
  PIGF cycle 1 day 15 | 81.6 [51.5 to 112]
  VEGF cycle 2 day 1 | 243.4 [136.1 to 418.1]
  PIGF cycle 2 day 1 | 68.8 [49.9 to 88]
  VEGF end of study (eos) | 184.3 [62.9 to 311.6]
  PIGF end of study (eos) | 53.5 [32.4 to 100]
Statistical Analysis 1: Comparison: Sorafenib & TRC105 in Hepatocellular CA; Test type: Non-Inferiority — Paired T-test. Two tailed; p < 0.05, Wilcoxon signed rank test

17. Secondary Outcome: Changes in Biomarker Cluster of Differentiation 105 (CD105)
Description: Blood samples were collected and analyzed by the enzyme-linked immunosorbent assay (ELISA). Serum samples were measured using a validated ELISA with a lower limit of quantification (LLOQ) of 200 ng/ml. Soluble endoglin was only assessed in patient samples without detectable TRC105 concentrations.
Time Frame: Cycle 1 day 1, cycle 1 day 15, cycle 2 day 1, or end of study (eos), an average of 12 weeks
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Sorafenib & TRC105 in Hepatocellular CA
Number analyzed (Participants) | 25
ng/ml
  Cycel 1 Day 1 | 27.5 [22.9 to 36]
  Cycle 1 Day 15 | 60.4 [41 to 78.5]
  Cycel 2 day 1 | 64.5 [51.4 to 87.3]
  End of study (eos) | 66.6 [31.5 to 86.4]
Statistical Analysis 1: Comparison: Sorafenib & TRC105 in Hepatocellular CA; Test type: Non-Inferiority — Paired T-test. Two tailed; p < 0.0001, Wilcoxon signed rank test — Cycle 1 day 15 vs. cycle 1 day 1
Statistical Analysis 2: Comparison: Sorafenib & TRC105 in Hepatocellular CA; Test type: Non-Inferiority — Cycle 2 day 1 vs. cycle 1 day 1. Paired T-test. Two tailed; p < 0.0001, Wilcoxon signed rank test
Statistical Analysis 3: Comparison: Sorafenib & TRC105 in Hepatocellular CA; Test type: Non-Inferiority — eos (end of study) vs. cycle 1 day 1. Paired T-test. Two tailed; p = 0.0009, Wilcoxon signed rank test

18. Secondary Outcome: Percentage Signal Change in Response on Magnetic Resonance Imaging (MRI)
Description: The perfusion of tumors was evaluated and analysis of normalized signal intensity in unenhanced and enhanced MRIs at each time point with calculation of measured percentage of signal change to reflect tumor vascularity. Signal change and signal intensity is defined as the Initial Area Under the Gd Curve measured over 60 seconds (IAUC60) and the Transport Constant (Ktrans) and the difference in these values relative to baseline.
Time Frame: Baseline and Cycle 1 Day 2 and Cycle 2 Day 1, an average of 12 weeks
Population: This analysis was not done as magnetic resonance imaging (MRI) scans not performed as planned.
Arm/Group | Sorafenib & TRC105 in Hepatocellular CA
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 4 years and 10.5 months
Description: 16 deaths are not included in the serious adverse event table because this study was originally not under the death related to disease serous adverse event. The deaths were reported in the continuing reviews.
Arm/Group | Sorafenib & TRC105 in Hepatocellular CA
All-Cause Mortality (participants affected / at risk) | 16/27
Serious Adverse Events (participants affected / at risk) | 11/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib & TRC105 in Hepatocellular CA (N=27)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (2)
Hypotension (Vascular disorders) | 1 (1)
Infusion related reaction (General disorders) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
Lipase increased (Investigations) | 1 (3)
Lung infection (Infections and infestations) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Serum amylase increased (Investigations) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib & TRC105 in Hepatocellular CA (N=27)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 12 (27)
Alanine aminotransferase increased (Investigations) | 16 (45)
Alkaline phosphatase increased (Investigations) | 17 (41)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5)
Anemia (Blood and lymphatic system disorders) | 21 (62)
Anorexia (Metabolism and nutrition disorders) | 8 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 4 (5)
Aspartate aminotransferase increased (Investigations) | 18 (62)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 17 (60)
Bronchial infection (Infections and infestations) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Cold sensitivity (Nervous system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Creatinine increased (Investigations) | 6 (10)
Dehydration (Metabolism and nutrition disorders) | 4 (5)
Diarrhea (Gastrointestinal disorders) | 13 (31)
Dizziness (Nervous system disorders) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4)
Dysgeusia (Nervous system disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Edema limbs (General disorders) | 5 (8)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Enterocolitis infectious (Gastrointestinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 17 (36)
Eye disorders - Other, Bleeding; Puffy eyelids (Eye disorders) | 2 (2)
Fatigue (General disorders) | 17 (25)
Fever (General disorders) | 8 (9)
Fibrinogen decreased (Investigations) | 1 (2)
Flu like symptoms (General disorders) | 2 (2)
Flushing (Vascular disorders) | 3 (3)
Gait disturbance (General disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 3 (6) — Gingival hemorrhage; Gum bleeding; Gums reddened; Indigestion-chest area; virus
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Gastroparesis (Gastrointestinal disorders) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) — Weakness
Gingival pain (Gastrointestinal disorders) | 4 (4)
Headache (Nervous system disorders) | 17 (39)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hot flashes (Vascular disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 6 (7)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (5)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (4)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 6 (12)
Hyperuricemia (Metabolism and nutrition disorders) | 6 (17)
Hypoalbuminemia (Metabolism and nutrition disorders) | 20 (53)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 5 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 7 (14)
Hyponatremia (Metabolism and nutrition disorders) | 13 (28)
Hypophosphatemia (Metabolism and nutrition disorders) | 22 (56)
Hypotension (Vascular disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 5 (10) — Infection-tooth; Infection-wisdom tooth; Respiratory infection symptoms; Sinusitis; Thrush; Urinary infection; Urinary tract infection; Thrush infection
Infusion related reaction (General disorders) | 8 (11)
Insomnia (Psychiatric disorders) | 3 (3)
Lipase increased (Investigations) | 1 (1)
Lung infection (Infections and infestations) | 1 (2)
Lymphocyte count decreased (Investigations) | 17 (50)
Malaise (General disorders) | 2 (6)
Mucositis oral (Gastrointestinal disorders) | 4 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Nausea (Gastrointestinal disorders) | 13 (26)
Neutrophil count decreased (Investigations) | 6 (11)
Oral hemorrhage (Gastrointestinal disorders) | 3 (4)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 18 (47)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (6)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 10 (27)
Periodontal disease (Gastrointestinal disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Platelet count decreased (Investigations) | 10 (23)
Proteinuria (Renal and urinary disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5)
Radiculitis (Nervous system disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 14 (52)
Rectal fistula (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 (1) — Vaginal heat
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Seasonal allergies
Rhinitis infective (Infections and infestations) | 1 (1)
Serum amylase increased (Investigations) | 12 (31)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 (8) — Hand Foot Syndrome
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (2)
Somnolence (Nervous system disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 2 (2)
Upper respiratory infection (Infections and infestations) | 3 (3)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Vomiting (Gastrointestinal disorders) | 6 (12)
Weight loss (Investigations) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
White blood cell decreased (Investigations) | 10 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-07-07): https://cdn.clinicaltrials.gov/large-docs/58/NCT01306058/Prot_SAP_ICF_000.pdf